CLINICAL TRIAL: NCT04059744
Title: Experience and Technology Acceptance of Older Adults Towards a Gamified Rehabilitative Device Prototype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Eng Chan Neoh, Senior Physiotherapist, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/01111
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Convenience sampling will be used. Participants will be recruited through email.
  Participants will be number-coded.Participants will be guided to put on the Fun-Knee sleeve. They will perform 3 repetitions of maximal knee flexion and maximal knee extension. A delegated study team member will teach the participant to use the mobile game application that is preloaded on a provided smartphone. Thereafter, they will be given time to complete two games at their own pace, inside a quiet, conducive room. After their trial use of the Fun-Knee prototype, participants will be asked to complete a survey on their experience and impression of Fun-Knee. Following that, a few open-ended questions will be asked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Device: Fun-Knee Portable and low cost sensors are used in the Smart Knee Sleeve. The sensor system is composed of two inclinometers and one Bluetooth transmitter.
  Fun Knee™ contains total knee replacement exercises that are gamified and supported on mobile device running on Android or iOS platforms. The mobile apps is able to capture the angle a and position data from the two inclinometers on smart knee sleeve.The free-sized knee sleeve prototypes are purchased and assembled by our collaborating vendor.
  Interventions: Device: Fun-Knee

INTERVENTIONS:
Device: Fun-Knee — Portable and low cost sensors are used in the Smart Knee Sleeve. The sensor system is composed of two inclinometers and one Bluetooth transmitter.
  Fun Knee™ contains total knee replacement exercises that are gamified and supported on mobile device running on Android or iOS platforms. The mobile apps is able to capture the angle a and position data from the two inclinometers on smart knee sleeve.The free-sized knee sleeve prototypes are purchased and assembled by our collaborating vendor.

SUMMARY:
Title: Older adults' experience and acceptance of a 'gamified' rehabilitative device for Total Knee Arthroplasty Background: Total Knee Arthroplasty (TKA) is a common surgical procedure. Good post-operative rehabilitation is needed for successful functional recovery. Patients in our institution demonstrated reduced exercise compliance and accuracy during early post-operative rehabilitation. Root cause analysis identified 'reduced feedback', 'reduced care continuity' and 'lack of engagement' to be key contributing factors. Yet, healthcare resource limitations necessitate new ways of care continuation and patient activation. In response, Fun-Knee™, an app-based innovation was created. Using 'gamification' of rehabilitative exercises, Fun-Knee™ guides and tracks rehabilitation from post-surgery to after hospital discharge, till outpatient physiotherapy review. The experience and opinions of older adults towards such 'gamified' rehabilitative technology is unknown.

Purpose: This feasibility study aims to evaluate and develop Fun-Knee™, a novel, app-based rehabilitation device that 'gamifies' post-TKA exercises to improve exercise compliance, effectiveness, and patient activation. Our prototype of Fun-Knee™ was introduced to two cohorts of healthy older adults. Users' experience with hardware and software components of Fun-Knee™, and their acceptance of Fun-Knee™ for rehabilitation were surveyed. Feedback from the first cohort guided prototype refinement. User experience was re-evaluated in the second cohort.

Methods: Community-dwelling adults with no knee pain, 50 years old and above were recruited if they met inclusion criteria. Participants were introduced to two 'gamified' exercises within Fun-Knee™ with standardised instructions. They were instructed to complete one round of the two games at their own time. Thereafter, a survey consisting of quantitative responses was administered. Statistical analysis were performed using Stata (version 13.1, College Station, TX: StataCorp LP), Fisher's exact tests were performed 2-sided at the 5% significance level. Qualitative feedback was obtained during individual interview. Suggestions for hardware or software refinements to Fun-Knee™ were collated and implemented. The above process was repeated for the second cohort of participants, using the latest version of Fun-Knee™.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact (able to follow 3 step commands), community dwelling adults who are 50 years old and above. Not currently attending physiotherapy for knee pain.

Exclusion Criteria:

* Lower limb skin sensitivity, lower limb sensory impairment, open wounds or broken skin, severe vision or hearing impairment, presence of knee pain above 3/10 on numerical rating scale and being English/ Chinese illiterate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
survey | through study completion, an average of 3 months
  A survey on their experience and impression of Fun-Knee. Following that, a few open-ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Eng Chuan Neoh, Principal Investigator — Senior Physiotherapist
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No